CLINICAL TRIAL: NCT03699423
Title: Evaluation of Two-week Effects of 0.01%, 0.02% and 0.03% Atropine Eye Drops on Children Eyes With Myopia
Brief Title: Effects of Low Concentration Atropine on Pupillary Size and Accommodative Amplitude
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hai Yen Eye Care (Industry)
Collaborators: Brien Holden Vision (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CS_AS_18_07
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Myopia
Keywords: myopia control; low concentration atropine eye drops; anti-muscarinic receptors; pupil size; accommodative amplitude
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study treatments will be labelled as A, B and C by one of the team member who does not involve in the assessment and follow-up. The masked study products will then be sent to the study coordinator to dispense
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.01% atropine eye drops (Active Comparator): Participants will receive one drop per eye every night for two weeks
  Interventions: Drug: 0.01% atropine eye drops
- 0.02% atropine eye drops (Active Comparator): Participants will receive one drop per eye every night for two weeks
  Interventions: Drug: 0.02% atropine eye drops
- 0.03% atropine eye drops (Active Comparator): Participants will receive one drop per eye every night for two weeks
  Interventions: Drug: 0.03% atropine eye drops

INTERVENTIONS:
Drug: 0.01% atropine eye drops — 0.01% atropine sulphate
  Arms: 0.01% atropine eye drops
Drug: 0.02% atropine eye drops — 0.02% atropine sulphate
  Arms: 0.02% atropine eye drops
Drug: 0.03% atropine eye drops — 0.03% atropine sulphate
  Arms: 0.03% atropine eye drops

SUMMARY:
To assess the two-week ocular responses, especially on pupillary size and accommodative amplitude, of nightly application of 0.01% or 0.02% or 0.03% atropine eye drops in children with myopia who were randomized to use of three different low-concentration atropine eye drops

DETAILED DESCRIPTION:
Atropine was proven to be effective in controlling myopia progression. However, the most common side effects of the use of atropine eye drop are dilation of pupil and decrease of accommodation. The investigators wish to evaluate the ocular responses of three low concentration atropine eye drops, 0.01% or 0.02% or 0.03%, mainly on the pupillary size and accommodative responses in children aged between 6 to 12 years old over two-week usage.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and comprehend Vietnamese and having parents or legal guardians who give informed consent as demonstrated by signing a record of informed consent.
* Be between 6 and 12 years old, male or female.
* Willing to apply eye drops once nightly at bedtime for two weeks and follow the clinical trial visit schedule as directed by the Investigator.
* Willing to answer the questionnaire about subjective measurements
* Have ocular findings deemed to be normal
* No contact lens wearing history
* Vision correctable to at least 20/25 or better in each eye with spectacles

Exclusion Criteria:

* Any pre-existing ocular irritation, injury or condition, including infection or disease.
* Any systemic disease that adversely affects ocular health e.g. diabetes, Graves disease, and auto-immune diseases such as ankylosing spondylitis, multiple sclerosis, Sjögrens syndrome and systemic lupus erythematosus. Conditions such as systemic hypertension and arthritis do not automatically exclude prospective participants.
* Use of or a need for concurrent category S3 and above ocular medication at enrolment and/or during the clinical trial.
* Use of or a need for any systemic medication or topical medications which may alter normal ocular findings / are known to affect a participant's ocular health / physiology or contact lens performance either in an adverse or beneficial manner at enrolment and/or during the clinical trial.

NB: Systemic antihistamines are allowed on an "as needed basis", provided they are not used prophylactically during the trial and at least 24 hours before the clinical trial product is used.

* History of eye surgery
* History of use of any myopia control interventions such as Orthokeratology, Rigid Permeable Contact Lenses Eye surgery within 12 weeks immediately prior to enrolment for this trial.
* Currently treated with other interventions for myopia control
* Contraindications to atropine such as pulmonary disease, heart conditions and ADHD
* Known allergy or intolerance to ingredients to atropine eye-drops and other derivatives of anti-muscarinic receptor agents.
* Currently enrolled in another clinical trial.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in pupillary diameter | at baseline, at three day and at two week
  Measure and compare the photopic and mesopic pupil size (milimeters) before and after instillation of eye drops
Change in accommodative amplitude | at baseline, at three day and at two week
  Measure and compare the accommodative amplitude (diopters) before and after instillation of eye drops

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology - An Sinh Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Background] Sankaridurg PR, Holden BA. Practical applications to modify and control the development of ametropia. Eye (Lond). 2014 Feb;28(2):134-41. doi: 10.1038/eye.2013.255. Epub 2013 Dec 6. PMID 24310242
- [Background] Huang J, Wen D, Wang Q, McAlinden C, Flitcroft I, Chen H, Saw SM, Chen H, Bao F, Zhao Y, Hu L, Li X, Gao R, Lu W, Du Y, Jinag Z, Yu A, Lian H, Jiang Q, Yu Y, Qu J. Efficacy Comparison of 16 Interventions for Myopia Control in Children: A Network Meta-analysis. Ophthalmology. 2016 Apr;123(4):697-708. doi: 10.1016/j.ophtha.2015.11.010. Epub 2016 Jan 27. PMID 26826749
- [Background] Polling JR, Kok RG, Tideman JW, Meskat B, Klaver CC. Effectiveness study of atropine for progressive myopia in Europeans. Eye (Lond). 2016 Jul;30(7):998-1004. doi: 10.1038/eye.2016.78. Epub 2016 Apr 22. PMID 27101751
- [Background] Chia A, Lu QS, Tan D. Five-Year Clinical Trial on Atropine for the Treatment of Myopia 2: Myopia Control with Atropine 0.01% Eyedrops. Ophthalmology. 2016 Feb;123(2):391-399. doi: 10.1016/j.ophtha.2015.07.004. Epub 2015 Aug 11. PMID 26271839
- [Background] Cooper J, Eisenberg N, Schulman E, Wang FM. Maximum atropine dose without clinical signs or symptoms. Optom Vis Sci. 2013 Dec;90(12):1467-72. doi: 10.1097/OPX.0000000000000037. PMID 24076540
- [Derived] Tran HDM, Ha TTX, Tran YH, Coroneo M, Tran TD, Truong TU, Sankaridurg P. Impact of Various Concentrations of Low-Dose Atropine on Pupillary Diameter and Accommodative Amplitude in Children with Myopia. J Ocul Pharmacol Ther. 2024 May;40(4):232-239. doi: 10.1089/jop.2023.0173. Epub 2024 Apr 15. PMID 38621178